CLINICAL TRIAL: NCT02922946
Title: A 2-Stage, Open-Label, Randomized, Single-Dose, Crossover Study to Determine the Effect of the Timing of a Meal on the Pharmacokinetics of Entinostat in Healthy Adult Subjects
Brief Title: Study to Determine the Effect of the Timing of a Meal on the Pharmacokinetics of Entinostat
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Syndax Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SNDX-275-0180
Record Dates: First submitted 2016-09-30; First posted 2016-10-04 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Volunteers; Healthy Volunteers; Human Volunteers; Normal Volunteers
Keywords: entinostat; Histone Deacetylase Inhibitor; HDAC
MeSH Terms: interventions — entinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Entinostat 5mg in 2-Way Crossover (Experimental): Treatment A: 5mg entinostat following an overnight fast and followed by a 4-hour fast.
  Treatment B: 5mg entinostat 2 hours after the completion of a meal and followed by a 1-hour fast.
  Interventions: Drug: Entinostat
- Entinostat 5mg in 3-Way Crossover (Experimental): Treatment C: 5mg entinostat following an overnight fast and followed by a 4-hour fast.
  Treatment D: 5mg entinostat following an overnight fast and 1 hour before the start of a meal.
  Treatment E: 5mg entinostat 2 hours after the completion of a meal and followed by a 4-hour fast.
  Interventions: Drug: Entinostat

INTERVENTIONS:
Drug: Entinostat — HDAC (histone deacetylase) inhibitor
  Other Names: SNDX-275; MS-275

SUMMARY:
The objectives of this study are to evaluate the effect of the timing of a moderate-fat meal on the single dose pharmacokinetics of entinostat and to evaluate the safety and tolerability of entinostat under fed and fasting conditions in healthy adult subjects.

DETAILED DESCRIPTION:
This is a 2-stage food effect (timing of the meal) study. A total of 48 subjects will be dosed if Stage 2 is conducted.

Stage 1 will be conducted as an open-label, randomized, 2-way crossover study. On Day 1 of each period, subjects will receive a single, oral dose of entinostat under fasting or fed conditions.

If preliminary results in Stage 1 indicate that the timing of a meal exhibits significant effect on the bioavailability of entinostat, then Stage 2 will be conducted which will investigate the effect of a meal either before or after dosing of entinostat on entinostat PK.

Stage 2 will be conducted as an open-label, randomized, 3-way crossover study. On Day 1 of each period, subjects will receive a single, oral dose of entinostat under fasting or fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 19-55 years of age at screening.
* Continuous non-smoker who has not used nicotine-containing products for at least 3 months prior to first dose and throughout the study.
* Body mass index of ≥ 18.5 at screening.
* Medically healthy with no significant medical history, physical examination, laboratory values, vital signs, or ECGs. Liver function tests and serum bilirubin must be ≤ the upper limit of normal. Platelets, hemoglobin, and hematocrit must be > the lower limit of normal at screening.
* Females of non-childbearing potential must have undergone sterilization procedures as noted in protocol at least 6 months prior to dose.
* Non-vasectomized male subjects must agree to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days beyond dose of study drug.
* Male subjects must agree not to donate sperm from the first dose until 90 days beyond dose of study drug.
* Understands the study procedures in the informed consent form and be willing and able to comply with the protocol.

Exclusion Criteria:

* Mentally or legally incapacitated or has significant emotional problems at screening or expected during the conduct of the study.
* History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee.
* History of illness that might confound the results of the study or poses an additional risk to the subject by their participation in the study in the opinion of the PI or designee.
* History of presence of alcoholism or drug abuse within the past 2 years prior to dose.
* History or presence of clinically significant cancer, cardiovascular disorders, acute or chronic gastrointestinal conditions in the opinion of the PI.
* Females of childbearing potential.
* Females with a positive pregnancy test or lactating.
* Positive urine drug or alcohol results are screening or each check-in.
* Positive urine cotinine at screening.
* Positive results are screening for HIV, hepatitis B surface antigen, or hepatitis C virus
* Seated blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg at screening.
* Seated heart rate lower than 40 bpm or higher than 99 bpm at screening.
* QTcB interval (correction value of the interval between the Q and T waves on the ECG tracing using the Bazett Correction Formula) > 460 msec for males or > 480 msec for females or has ECG findings deemed abnormal by the PI or designee.
* Estimated creatinine clearance < 90 mL/min at screening.
* Unable to refrain from or anticipates the use of any prescription or non-prescription medications and any drugs known to be significant inhibitors or CYP (Cytochromes 450) enzymes and/or P-gp.
* Has been on a diet incompatible with the on-study diet within 28 days prior to dose and throughout the study in the opinion of the PI or designee.
* Is lactose intolerant.
* Donation of blood or significant blood loss within 56 days prior to dose.
* Plasma donation within 7 days prior to dose.
* Participation in another clinical study 28 days prior to dose.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2016-10-11 (Actual); Primary Completion 2017-05-20 (Actual); Study Completion 2017-06-26 (Actual)

PRIMARY OUTCOMES:
AUC0-t (area under the concentration-time curve, from time 0 to the last observed non-zero concentration (t) for entinostat under fed and fasting conditions | Pre-dose through Day 22
AUC0-inf (area under the concentration-time curve, from time 0 extrapolated to infinity) for entinostat under fed and fasting conditions | Pre-dose through Day 22
Cmax (maximum observed concentration) of entinostat under fed and fasting conditions | Pre-dose through Day 22
AUC%extrap (percent of AUC0-inf extrapolated) of entinostat under fed and fasting conditions | Pre-dose through Day 22
Tmax (time to reach maximum observed concentration) of entinostat under fed and fasted conditions | Pre-dose through Day 22
Kel (apparent terminal elimination rate constant) of entinostat under fed and fasted conditions | Pre-dose through Day 22
T1/2 (apparent terminal elimination half-life) of entinostat under fed and fasted conditions | Pre-dose through Day 22
Changes from baseline in physical exam | Baseline through Day 1
Changes from baseline in vital signs | Baseline through Day 22
Changes from baseline in ECG results | Baseline through Day 22
Changes from baseline in adverse events | Baseline through 14 days after last sample collection
Changes from baseline in clinical laboratory tests | Baseline through Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Laura Sterling, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No
Data will be reviewed throughout the study by the sponsor, clinical research organization assisting with serious adverse event management, and routine monitoring to safeguard the interests of the trial subjects and to assess the safety of the interventions administered during the trial.